CLINICAL TRIAL: NCT03949088
Title: Integrated Strategies to Prevent Intradialytic Hypotension: a Prospective Randomized Cross-over Trial in Hypotension-prone Hemodialysis Patients (The DialHypot Study)
Brief Title: Integrated Strategies to Prevent Intradialytic Hypotension (The DialHypot Study)
Acronym: DialHypot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Parma (Other)
Responsible Party: Principal Investigator, Enrico Fiaccadori, University Professor, University of Parma
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: DialHypot
Record Dates: First submitted 2019-05-07; First posted 2019-05-14 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Hypotension During Dialysis; Dialysis Hypotension
Keywords: Intradialytic hypotension (IDH); Ultrafiltration (UF) profiling; Sodium (Na) profiling; Hemodialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Linear descending UF profile (Experimental): 2-step descending Na profile, linear descending UF profile 3 weeks (9 sessions)
  Interventions: Other: UF and Na profiling
- Run-in & washout phases (Experimental): constant Na concentration, constant UF rate 3 weeks (6+3 sessions)
  Interventions: Other: UF and Na profiling
- Ascending/descending UF profile (Experimental): 2-step descending Na profile, ascending/descending UF profile 3 weeks (9 sessions)
  Interventions: Other: UF and Na profiling

INTERVENTIONS:
Other: UF and Na profiling — Modulation of UF and dialysate sodium

SUMMARY:
The present study is aimed at comparing different strategies of UF profiling, dialysate sodium individualization and sodium profiling (even combining one with the other) and at evaluating the effectiveness of a new UF profile which has an ascending/descending shape. The goal of the study is to provide better dialysis tolerance and lower rates of intradialytic hypotensive events by the application of this UF profile design in combination with a neutral sodium balance.

DETAILED DESCRIPTION:
This is a prospective, randomized, crossover trial. The study will be performed in 2 phases. Each phase will be divided in several sub-phases (see "4.1 Study phases"). Phase 1 will consist of 9 weeks of treatment (27 HD sessions) for each patient; phase 2 will consist of 11 weeks of treatment (33 HD sessions) for each patient. Each subject will be used as his/her own control. Dry weight, anti-hypertensive medications and dialysis parameters will not be modified during the study phases, except for UF rate and dialysate sodium concentration.

Study phases

1 - First phase: validation of the new UF profile with a standard dialysate sodium concentration

1. run-in: constant Na concentration, constant UF rate - 2 weeks (6 sessions)
2. 2-step descending Na profile, linear descending UF profile - 3 weeks (9 sessions)
3. washout: constant Na concentration, constant UF rate - 1 week (3 sessions)
4. 2-step descending Na profile, ascending/descending UF profile - 3 weeks (9 sessions)

2 - Second phase: combination of UF profiles and individualized dialysate sodium concentration

1. run-in: standard constant Na concentration, constant UF rate - 2 weeks (6 sessions)
2. individualized constant Na concentration, constant UF rate - 2 weeks (6 sessions)
3. individualized 2-step Na profile, linear descending UF profile - 3 weeks (9 sessions)
4. washout: individualized constant Na profile, constant UF rate - 1 week (3 sessions)
5. individualized 2-step Na profile, ascending/descending UF profile - 3 weeks (9 sessions)

In phase 1 patients will be randomly assigned to one of the following sequences:

* (1), (2), (3), (4)
* (1), (4), (3), (2)

In phase 2 patients will be randomly assigned to one of the following sequences:

* (1), (2), (3), (4), (5)
* (1), (2), (5), (4), (3) Patients who will be included in phase 1 will undergo at least a 2-week washout period before entering phase 2. During these 2 weeks dry weight and anti-hypertensive therapy may be re-evaluated and re-assessed.

Dialysis prescription

Every patient will undergo a standard HD with the following prescription:

* blood flow: individualized from 250 to 350 mL/min (this value will be established for each patient at the beginning of the run-in phase on the basis of previous evaluations and maintained unchanged for the whole duration of the study)
* dialysate flow: 500 mL/min
* dialysate composition: HCO3- 34 mmol/L, K+ 3 mmol/L, Ca2+ 1.25 mmol/L, Mg2+ 0.5 mmol/L, Cl- 111.5 mmol/L, acetate 3.0 mmol/L, glucose 1 g/L
* dialysate temperature: 36°C
* HD session duration: 4 hours
* during each dialysis session patients will be allowed to drink an amount of maximum 150 mL of water, tea or coffee and they will be allowed to eat a snack

UF profiles

* "linear descending" UF profile: this profile provides a constantly decreasing UF rate during dialysis, starting at a UF rate 1.33 fold the average UF rate (33,25% of total UF rate)
* "ascending/descending" UF profile: this profile can be divided in 2 different phases. The first one includes 3 ascending steps during the first hour of treatment, each step lasting 20 minutes (during the 1st step UF rate is set at 15% of total UF rate, during 2nd step at 25% of total UF rate, during 3rd step at 35% of total UF rate). During the following 3 hours UF rate is shaped as a linear descending UF profile, with a constantly decreasing UF rate, starting at a UF rate 1.33 fold the average UF rate (33,25% of total UF rate)

Dialysate sodium

1. - First phase

   * "standard" concentration: the investigators will consider as "standard" a dialysate sodium concentration of 140 mmol/L, which is the concentration usually prescribed in our dialysis facility
   * dialysate sodium profile will be shaped as a descending 2-step ramping, each step consisting of half the total treatment duration (2 hours), with a 6 mmol/L difference between the concentrations defined for each of the two steps. Considering a monocompartimental model with variable dialysate sodium, the profile will be set on the basis of an "equivalent sodium". This value will correspond to the dialysate sodium concentration expected to produce the same diffusive balance that a fixed standard concentration (140 mmol/L) would provide: 144 mmol/L for the first 2 hours, 138 mmol/L for the last 2 hours
2. - Second phase

   * "individualized" concentration: for each patient dialysate sodium concentration will be established on the basis of the mean of the sodium plasma values measured through pre-HD sampling during the run-in phase (2 repeated measurements before each HD session, for a total of 12 values for each patient). Plasma values will be obtained through a direct potentiometry analysis. Dialysate sodium concentration will be set at the patient's average plasma sodium concentration
   * dialysate sodium profile will be shaped as a descending 2-step ramping, each step consisting of half the total treatment duration (2 hours), with a 6 mmol/L difference between the concentrations set for each of the two steps. Considering a monocompartimental model with variable dialysate sodium, the profile will be set on the basis of an "equivalent sodium". This value will correspond to the dialysate sodium concentration expected to produce the same diffusive balance that a fixed individualized concentration (equal to the patient's average plasma sodium concentration) would provide: "average + 4" mmol/L for the first 2 hours, "average - 2" mmol/L for the last 2 hours

Definition of "dry weight", "UF volume" and "interdialytic weight gain"

* dry weight will be estimated through standard clinical criteria
* total UF volume (net fluid to be removed) will be calculated before each session as the difference between patient's weight and his/her dry weight. A limit of 12.5 mL/kg/h will be considered as maximal total UF volume
* IDGW will be calculated as the difference between patient's weight at the beginning of dialysis and the weight registered at the end of the previous session UF and IDGW will be respectively corrected for pre-HD weight (UF %) and dry weight (IDWG %), thus obtaining measures that will be more relevant to each specific patient.

Primary outcome and definition of "intradialytic hypotension"

The primary outcome will be the incidence of intradialytic hypotensive episodes. Hypotensive events and symptoms (headache, cramps, nausea and vomiting) will be recorded and analyzed as both number of occurrences and time of occurrence from the beginning of the HD session. IDH will be defined as follows:

* "symptomatic IDH": decrease in SBP ≥ 20 mmHg or in MAP ≥ 10 mmHg associated with symptoms (KDIGO definition)
* "asymptomatic IDH": drop in BP (SBP ≥ 20 mmHg or MAP ≥ 10 mmHg) within a 20 minutes interval, regardless of symptoms
* for patients whose SBP is < 100 mmHg at the beginning of treatment, the investigators will consider as IDH any decrease of SBP ≥ 10%

Interventions in case of hypotensive events

* Trendelenburg position
* temporary stop of UF (10 minutes), then restarted at a UF rate equal to "total UF - 100 mL"
* online infusion of 150 mL of saline solution
* discontinuation of the session

BV monitoring Relative blood volume will be evaluated through the BVM system integrated in the dialysis machine. RBV will be recorded every 10 minutes.

Other outcome measurements

* pre-, intra- (after every hour of treatment) and post-HD plasma sodium levels will be determined by direct potentiometry
* blood pressure and heart rate will be recorded every 20 minutes, or more frequently if needed for clinical necessities, by machine-integrated BPM
* achievement of UF will be considered as:

  * achievement of dry weight: % target UFDW = UF vol / (preHD weight - dry weight) x 100
  * IDWG removal: % target UFWG = UF vol / IDWG x 100
* "UF failure" will be defined as % target UFDW < 70%
* "session failure" will occur when treatment will have to be discontinued before 75% of the prescribed time (before 3 hours of treatment)
* Kt/V will be estimated through the system integrated in the machine (total body water calculated using Watson's equation)

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* age ≥ 18 years
* thrice weekly HD regimen for more than 6 months
* "hypotension-prone patients": ≥ 3 episodes of IDH in the month preceding the run-in phase of the study

Exclusion Criteria:

* IDWG < 1.4% of dry weight (corresponding to < 1 kg in a 70-kg person)
* twice weekly HD regimen
* residual daily urine output > 300 mL
* active acute disease or hospitalization in the 8 weeks preceding the run-in phase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of intradialytic hypotensive episodes (number of episodes within every HD session and time interval from HD start) | Within each dialysis session from the time of enrolment to the end of each study phase (9-11 weeks)
  Hypotensive events and symptoms (headache, cramps, nausea and vomiting) will be recorded and analyzed as both number of occurrences and time of occurrence from the beginning of the HD session.
  IDH will be defined as follows:
  * "symptomatic IDH": decrease in SBP ≥ 20 mmHg or in MAP ≥ 10 mmHg associated with symptoms (KDIGO definition)
  * "asymptomatic IDH": drop in BP (SBP ≥ 20 mmHg or MAP ≥ 10 mmHg) within a 20 minutes interval, regardless of symptoms
  * for patients whose SBP is < 100 mmHg at the beginning of treatment, the investigators will consider as IDH any decrease of SBP ≥ 10%

SECONDARY OUTCOMES:
Achievement of UF | Within each dialysis session from the time of enrolment to the end of each study phase (9-11 weeks)
  * achievement of dry weight: % target UFDW = UF vol / (preHD weight - dry weight) x 100
  * IDWG removal: % target UFWG = UF vol / IDWG x 100
  "UF failure" will be defined as % target UFDW < 70% "session failure" will occur when treatment will have to be discontinued before 75% of the prescribed time (before 3 hours of treatment)
Dialysis dose | Within each dialysis session from the time of enrolment to the end of each study phase (9-11 weeks)
  Kt/V: estimated through the system integrated in the machine (total body water calculated using Watson's equation)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Parma - UO Nefrologia AOU, Parma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peyronel F, Parenti E, Fenaroli P, Benigno GD, Rossi GM, Maggiore U, Fiaccadori E. Integrated strategies to prevent intradialytic hypotension: research protocol of the DialHypot study, a prospective randomised clinical trial in hypotension-prone haemodialysis patients. BMJ Open. 2020 Jul 8;10(7):e036893. doi: 10.1136/bmjopen-2020-036893. PMID 32641335